CLINICAL TRIAL: NCT02356029
Title: The REAppropriate Study: Perception of Inappropriate CPR: a Multicenter International Cross-sectional Survey
Brief Title: Perception of Inappropriate CPR: a Multicenter International Cross-sectional Survey
Acronym: REAppropriate
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B670201422126
Record Dates: First submitted 2015-01-14; First posted 2015-02-05 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Cardiopulmonary Arrest
Keywords: Cardiopulmonary Arrest; Emergency Medical Services; Medical Futility; Decision Making; Emotional Stress; Burnout, Professional
MeSH Terms: conditions — Heart Arrest; Stress, Psychological; Burnout, Professional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EMS Healthcare Providers: Healthcare Providers working in Emergency Medical Services and directly involved in treatment of cardiac arrest patients (out-of-hospital or in the Emergency Department)

SUMMARY:
The primary objective of this study is to determine how often cardiopulmonary resuscitation (CPR) is perceived as inappropriate by Healthcare Providers (HCPs) working in prehospital Ambulance Services and Emergency Departments. Perception of inappropriate CPR is defined as resuscitation efforts perceived by HCPs as disproportionate to the expected prognosis of the patient in terms of survival or quality of life.

When a HCP perceives CPR as inappropriate, this may cause moral and emotional distress. This perception may be modulated by the personal background and professional role of the HCP, but also by his/her working conditions. Apart from the workload, the resulting distress can be influenced by the way non-technical skills are developed within the team and the ethical environment in which the HCP functions. Frequent exposure to similar patient care situations and/or a professional environment not acknowledging the distress may lead to deficient coping mechanisms and accumulation of moral distress. This may be associated with job leave, burnout and a decreased quality of patient care. Acute distress may also influence the quality of care provided to actual and future patients.

Secondary objectives of the study are to evaluate whether perceived inappropriateness of CPR is not only associated with patient related factors but also with personal characteristics and work related factors. Potential consequences for HCP's like moral distress and intentional job leave will be assessed.

DETAILED DESCRIPTION:
The REAppropriate study is an international multicentric cross-sectional survey exploring perception of inappropriateness of CPR.

Objectives:

The primary objective of this study is to determine the prevalence of perceived inappropriateness of CPR (PICPR) of the last resuscitation performed out-of-hospital or in the Emergency Department (ED) by Healthcare Providers (HCP) working in prehospital Ambulance Services and EDs. PICPR is defined as resuscitation efforts perceived by HCPs as disproportionate to the expected prognosis of the patient in terms of survival or quality of life. Prevalence of PICPR is defined as the number of HCPs reporting PICPR in the last cardiac arrest situation they attended divided by the total number of surveyed HCPs.

Secondary objectives are to evaluate the hypothesis that PICPR is not only associated with patient related factors but also with personal characteristics and work related factors. Other objectives will be assessment of moral distress and intentional job leave.

In each participating country a National Coordinator is nominated by the Steering Committee. National Coordinators are selected because of their leading role in national or international scientific organisations related to Emergency Medicine and/or their teaching or research activities related to Emergency Medicine.

Each National Coordinator establishes a network of Local Investigators who coordinate study proceedings within EDs and Ambulance Services.

Study population:

The survey will focus on HCPs directly involved in treatment of cardiac arrest patients (out-of-hospital or in the ED): nurses, doctors, ED Technicians/Nurse Assistants and Emergency Medical Technicians(EMT)/Paramedics working in EDs and prehospital Ambulance Services active in the Emergency Medical Services system of the country. Hospitals in countries without established EDs but with a group of HCPs working inside the hospital and having as their daily duty the first care and stabilisation of patients arriving unplanned in the hospital are also eligible for participation in the study. The Local Investigator will clearly delineate this functional unit within the hospital thus determining the number of eligible HCPs within the center.

Survey:

Two electronic questionnaires will be used: one for the Local Investigator of the ED or Ambulance Service and one for the HCPs.

Questionnaire for Local Investigator: this questionnaire requests quantitative data on organisational issues like number of beds, ED or Ambulance Service activity, number of doctors, nurses, EMTs/Paramedics etc. and a few questions about resuscitation practice.

Questionnaire for HCPs: the HCPs are asked about their personal characteristics and educational background. There are questions about their working conditions, job strain and teamwork within their professional environment. Their opinion is asked about possible reasons and statements concerning perception of (in)appropriate resuscitation. Finally they are questioned about the last resuscitation they were involved in themselves (it will not be necessary for them to have the medical file available while answering these questions). The HCP is first asked an opinion about the (in)appropriateness of the intervention and the resulting amount of moral and emotional distress, should this be the case. This is followed by questions about the circumstances of the cardiac arrest and a query on the relative importance of patient related, situational and interprofessional items. Four level Likert items are used where appropriate. Interest level analysis will be incorporated in the questionnaire to assist in assessing nonresponse bias.

Completion of the questionnaire will take approximately 20 minutes. Participation is on a voluntary basis.

Translation of surveys:

A modified Brislin's model of translation will be used. The primary questionnaires are in English. Both questionnaires are being translated in additional languages (the so called target languages) using the following procedure:

1. The first step will be forward translation of the English questionnaire into the target language by two native speakers of the target language with a proficient knowledge of English and ideally with a background in the medical specialties covered by the topic of this research.
2. The second step is that a third person whose native language is the target language reviews the translated versions together with the translators of step 1 for grammatical style and comprehensibility without the English text (so this can be a monolingual person). The most appropriate forward translation is chosen.
3. When this has been achieved the third step is the back translation to the English language of the most appropriate forward translation by two different bilingual persons (ideally native English speaking with a proficient knowledge of the target language) who are blinded from the original English version. Again efforts are made that the back translators are professionally involved in the research field to improve the quality of the translation process. The two back translations are reviewed with a third person and the most appropriate back translation is chosen.
4. In the last and fourth step the Steering Committee compares the most appropriate back translation of both questionnaires with the original English version. If necessary, recommendations will be done for modifications.

Throughout this process regular interaction and feedback with the Steering Committee will further optimise the quality of the translation.

Information Technology:

All the data will be collected through the use of a website especially designed for this study. Normal web applications use HTTP (Hypertext Transfer Protocol) to transfer web pages between the web server and the web browser. In order to guarantee data safety a HTTPS website signed by a trusted certificate authority will be used for this project. All the transferred data are encrypted in these circumstances and can only be read by the web browser and the web server.

Ethics approval:

For the HCP no risk is associated with participation in the study since the survey is completely anonymous. Insight in medical files is unnecessary to complete the questionnaires.

The National Coordinator will submit the protocol to one or more national ethical committees according to the rules applied in his/her jurisdiction. Ethical approvals should be sent to the Steering Committee.

If necessary, written informed consent will be obtained from the participating HCPs. Otherwise, completion of the questionnaire by the HCP will be taken as evidence of consent to study participation. In countries where informed consent must be obtained, it is preferable that the informed consent is uniform for the whole country.

Centers are not allowed to retrieve and report data unless ethical approval or after reporting to the Steering Committee there is no requirement for ethical approval for their country.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare Provider working in Emergency Department or Ambulance Service directly involved in treatment of cardiac arrest patients

Exclusion Criteria:

* Healthcare Provider working in Emergency Department or Ambulance Service not directly involved in treatment of cardiac arrest patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The survey will focus on Healthcare Providers (HCPs) directly involved in treatment of cardiac arrest patients (out-of-hospital or in the Emergency Department (ED)): nurses, doctors, ED Technicians/Nurse Assistants and Emergency Medical Technicians(EMT)/Paramedics working in EDs and prehospital Ambulance Services active in the Emergency Medical Services system of the country. Hospitals in countries without established EDs but with a group of HCPs working inside the hospital and having as their daily duty the first care and stabilisation of patients arriving unplanned in the hospital are also eligible for participation in the study. The Local Investigator will clearly delineate this functional unit within the hospital thus determining the number of eligible HCPs within the center.
Sampling Method: Non-Probability Sample
Enrollment: 5882 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The number of Healthcare Providers (HCPs) reporting Perceived Inappropriateness of CPR (PICPR) in the last cardiac arrest situation attended divided by the total number of surveyed HCPs | 2 weeks

SECONDARY OUTCOMES:
Moral distress and intentional job leave associated with Perceived Inappropriateness of CPR (PICPR) | 2 weeks
  Moral distress defined as when one knows the right thing to do, but institutional constraints make it nearly impossible to pursue the right course of action

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M Druwé, MD, Principal Investigator — University Hospital, Ghent
Locations (5):
- Belgium (5):
  - UMC Sint-Pieter, Brussels
  - UVC Brugmann, Brussels
  - Groupe Jolimont, Haine-Saint-Paul
  - CHU Tivoli, La Louvière
  - CHU Vesale Charleroi, Montigny-le-Tilleul

REFERENCES:
- [Result] Marco CA, Bessman ES, Kelen GD. Ethical issues of cardiopulmonary resuscitation: comparison of emergency physician practices from 1995 to 2007. Acad Emerg Med. 2009 Mar;16(3):270-3. doi: 10.1111/j.1553-2712.2008.00348.x. Epub 2009 Jan 9. PMID 19183108
- [Result] Marco CA, Schears RM. Prehospital resuscitation practices: a survey of prehospital providers. J Emerg Med. 2003 Jan;24(1):101-6. doi: 10.1016/s0736-4679(02)00688-1. PMID 12554050
- [Result] Partridge RA, Virk A, Sayah A, Antosia R. Field experience with prehospital advance directives. Ann Emerg Med. 1998 Nov;32(5):589-93. doi: 10.1016/s0196-0644(98)70038-1. PMID 9795323
- [Derived] Druwe P, Monsieurs KG, Gagg J, Nakahara S, Cocchi MN, Elo G, van Schuppen H, Alpert EA, Truhlar A, Huybrechts SA, Mpotos N, Paal P, BjOrshol C, Xanthos T, Joly LM, Roessler M, Deasy C, Svavarsdottir H, Nurmi J, Owczuk R, Salmeron PP, Cimpoesu D, Fuenzalida PA, Raffay V, Steen J, Decruyenaere J, De Paepe P, Piers R, Benoit DD; REAPPROPRIATE study group. Impact of perceived inappropiate cardiopulmonary resuscitation on emergency clinicians' intention to leave the job: Results from a cross-sectional survey in 288 centres across 24 countries. Resuscitation. 2021 Jan;158:41-48. doi: 10.1016/j.resuscitation.2020.10.043. Epub 2020 Nov 20. PMID 33227397